CLINICAL TRIAL: NCT06972784
Title: Xiangya Cardiopulmonary Health and Disease Cohort
Acronym: XY-CPHDC
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022YFC3601001
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Function Tests，Heart Function Tests; Cardiopulmonary Function
Keywords: Respiratory function tests，Heart Function Tests，Cardiopulmonary function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort
- Prospective cohort

SUMMARY:
Xiangya Cardiopulmonary Health and Disease Cohort (XY-CPHDC) is a non-intervention study grounded in real-world data. It is designed as a bidrectional clinical cohort combined retrospective and prospective design, in order to evaluate cardiopulmonary function systematically and holistically, integrate physiology and medical theory, and explore the changing pattern of the cardiopulmonary under different health states. Cardiovascular System and Respiratory System are closely linked and interdependent physiological systems, and they play a vital role in maintaining normal life activities in the human body. Patients with cardiopulmonary disease often have conspicuous comorbidity characteristics, however, current measurements of cardiopulmonary function indicators are mostly limited to the assessments of single organ. This pattern of subspecialty care leads to deficiencies in the recognition of cardiopulmonary synergy dysfunction, and there is an urgent need for a more comprehensive and systematic approach to assessment. This study plans to construct a cardiopulmonary holistic assessment cohort, aiming at comprehensively and systematically reveal the intrinsic connection between the cardiopulmonary function in different scenarios, such as resting, exercise, and sleep, to deeply explore the core indicators of cardiopulmonary holistic function, to construct a joint stratification system of cardiopulmonary function, and to map cardiopulmonary comorbidity spectrum, so that they can accurately guide the diagnosis of the disease, the prognostic prediction and the intervention strategies.

DETAILED DESCRIPTION:
1.2.1 Study objective

1. Construct a cardiopulmonary holistic assessment cohort covering the full range of resting-exercise-sleep scenarios and encompassing non-cardiopulmonary disease-- cardiopulmonary hypofunction--cardiopulmonary disease populations in the longitudinal development of time.
2. Explore the core indicators related to cardiopulmonary hypofunction and disease risk, and construct a joint stratification system of cardiopulmonary function.
3. Map the cardiopulmonary comorbidity spectrum and describe its functional characteristics using the cardiopulmonary holistic assessment cohort, and analyze the impact of comorbidity patterns on patient's long-term prognosis and clinical outcomes.

1.2.2 Study type Bidirectional cohort design Retrospective cohort: Integrate historical hospital data(e.g., electronic medical records, imaging reports, cardiopulmonary function test records) and select the study population according to the inclusion and exclusion criteria.

Prospect cohort: patients from the retrospective cohort were screened to meet the study requirements and agreed to participate in subsequent studies for long-term follow-up(≥3years) and dynamic monitoring of cardiopulmonary function changes, 1.2.3 study content Building a cardiopulmonary cohort: build a full range of clinical cohort covering resting, exercise, and sleep scenarios with non-diseased, hypofunctional and cardiopulmonary disease populations, integrating retrospective data analysis and prospective follow-up monitoring to comprehensively reflect the cardiopulmonary performance of individuals in different physiological states, and laying the data foundation for subsequent analyses.

Constructing a joint stratification system for cardiopulmonary function: based on the data collected from the cardiopulmonary holistic assessment cohort, further in-depth feature extraction of cardiopulmonary function indicators is performed, and key indicators capable of predicting cardiopulmonary function decline and disease risk are screened out through data mining and dynamic monitoring, integrating the core indicators into a multidimensional risk indicator system, and stratifying patients by using a clustering method or based on a risk score, dividing low, medium and high risk groups, and realize the dynamic update of the stratification model.

Characterizing the cardiopulmonary comorbidity spectrum: Using the constructed cardiopulmonary cohort and the stratification system, we will deeply reveal the functional characteristics of cardiopulmonary comorbidity, analyze the functional changes and characteristics of patients with cardiopulmonary comorbidity in different scenarios (e.g., resting, exercising, or sleeping), and depict the characteristics of cardiopulmonary comorbidity spectrum; through the cardiopulmonary co-morbidity spectrum, we will deeply explore the interaction mechanism between the heart and the lungs in the progression of the disease, and analyze the impact of comorbidity on the prognosis and clinical outcomes of patients.

ELIGIBILITY:
I1 Inclusion and exclusion criteria for retrospective cohorts 1) Inclusion criteria:

1. Patients were either treated or hospitalized in the physical examination center, outpatient and emergency clinic in the Xiangya Hospital of Central South University from January 2010 to April 2025.
2. Completion of cardiac function (e.g., echocardiography) and pulmonary function (e.g., pulmonary function test) assessment, with an interval of no more than 1 year between the two.
3. Those who had complete clinical diagnostic and therapeutic information (e.g., medical history, medication records, laboratory test results, imaging reports) except for the cardiopulmonary function test report.

2)Exclusion criteria

1. Patients with complete loss of cardiopulmonary function test reports or key data (e.g., VO2peak, FEV1/FVC, LVEF).
2. Patients with loss of key clinical diagnostic and treatment data (e.g., medical history, medication records, laboratory test results).

2.1.2 Inclusion and exclusion criteria for prospective cohort

1）Inclusion criteria

1. Patients who have been included in the retrospective cohort.
2. Voluntarily signed informed consent form to participate in long-term follow-up for ≥3 years.
3. Able to complete the baseline assessment of the prospective cohort (including cardiopulmonary function retesting, questionnaires, etc.).
4. Stable conditions for follow-up (e.g., living in the local area, available valid contact information, no plans to move in the short term or go out for a long period of time).

2) Exclusion Criteria.

1. Patients who have been excluded from the retrospective cohort or for whom key data are missing.
2. With severe cognitive impairment, psychiatric disease or verbal communication disorder, unable to cooperate with follow-up and data collection.
3. Expected survival time <3 years (e.g., advanced malignancy, end-stage cardiopulmonary failure, etc.).
4. Incomplete cardiopulmonary function or other clinical data during the baseline assessment.
5. Those who plan to participate in other interventional clinical trials that may interfere with the assessment of cardiopulmonary function.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Xiangya Cardiopulmonary Health and Disease Cohort（ XY-CPHDC） is a bidirectional clinical cohort integrating retrospective and prospective designs to systematically evaluate cardiopulmonary functional synergy
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2035-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Death event | From participants agreed to participate in this study until the date of death from any or specific cause or the end of the study, whichever came first, assessed up to 10 years
  Death due to any cause or specific cause

SECONDARY OUTCOMES:
Life quality as measured by the 12-item short form health survey (SF-12). | Through study completion, an average of 3 years
  The seven situations of SF-12 include physical function, role limitations due to physical health or emotional problems, bodily pain, general health perceptions, vitality, and social function. The scoring criteria for the SF-12 scale is based on a percentage system, where higher scores indicate better quality of life
Hospitalization Costs | Through study completion, an average of 3 years
  Direct medical costs during hospitalization, including medication, diagnostic tests, therapeutic procedures, nursing care, and bed fees.Single admission: from admission to discharge; Multiple admissions: cumulative costs until study completion.Costs are inflation-adjusted and reported in RMB (USD equivalents provided for cross-regional comparisons when applicable).
Number of participants with cardiometabolic diseases or events | Through study completion, an average of 3 years
  The occurrence of cardiometabolic diseases or events (e.g. hypertension, heart failure, ACS and DM, etc.) are identified by self-report or their electronic health records and tests (e.g. blood pressure, blood glucose, lipids and hormone levels, echocardiogram, ECG etc.)
Number of participants with respiratory diseases or events | Through study completion, an average of 3 years
  The occurrence of respiratory diseases or events (e.g. COPD and asthma, or hospitalization due to exacerbation etc.) are identified by self-report or their electronic health records and tests (e.g. lung function test parameters, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University Affiliated, Changsha, Hunan, China